CLINICAL TRIAL: NCT04334980
Title: A Phase 1, Randomized, Observer-Blind, Placebo-Controlled Trial to Evaluate the Safety, Tolerability and Immunogenicity of the bacTRL-Spike Oral Candidate Vaccine for the Prevention of COVID-19 in Healthy Adults
Brief Title: Evaluating the Safety, Tolerability and Immunogenicity of bacTRL-Spike Vaccine for Prevention of COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symvivo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: bacTRL-Spike-1
Record Dates: First submitted 2020-03-31; First posted 2020-04-06 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- bacTRL-Spike (Experimental): * Group 1 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 1 billion colony forming units (cfu) of Bifidobacterium longum (B. longum);
  * Group 2 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 3 billion cfu of B. longum;
  * Group 3 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 10 billion cfu of B. longum;
  * Group 4 (n=3): Single Data and Safety Monitoring Board (DSMB)-defined dose of bacTRL-Spike among subjects 56 years of age and older.
  * Group 5 (n=12): DSMB-defined prime and boost doses of bacTRL-Spike delivered with a 28-day intervening interval.
  Interventions: Biological: bacTRL-Spike

INTERVENTIONS:
Biological: bacTRL-Spike — Each oral dose of bacTRL-Spike contains bacterial medium with either 1 billion (Group 1), 3 billion (Group 2) or 10 billion (Group 3) colony-forming-units of live Bifidobacterium longum, which has been engineered to deliver plasmids containing synthetic DNA encoding spike protein from SARS-CoV-2.

SUMMARY:
Protocol bacTRL-Spike-1 will be the first-in-human study of bacTRL-Spike, and the first-in-human use of orally delivered bacTRL. Each oral dose of bacTRL-Spike contains bacterial medium with either 1 billion (Group 1A), 3 billion (Group 2A) or 10 billion (Group 3A) colony-forming-units of live Bifidobacterium longum, which has been engineered to deliver plasmids containing synthetic DNA encoding spike protein from SARS-CoV-2.

DETAILED DESCRIPTION:
Protocol bacTRL-Spike-1 will be the first-in-human study of bacTRL-Spike, and the first-in-human use of orally delivered bacTRL. The trial is designed to evaluate the safety and tolerability of orally delivered bacTRL-Spike vaccine in healthy adults.

Total anticipated enrollment is n=24. The distribution of the sample size will be as follows:

* Group 1 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 1 billion colony forming units (cfu) of Bifidobacterium longum (B. longum);
* Group 2 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 3 billion cfu of B. longum;
* Group 3 (n=3; Sentinel +2): Single dose of bacTRL-Spike, equivalent to 10 billion cfu of B. longum;
* Group 4 (n=3): Single Data and Safety Monitoring Board (DSMB)-defined dose of bacTRL-Spike among subjects 56 years of age and older.
* Group 5 (n=12): DSMB-defined prime and boost doses of bacTRL-Spike delivered with a 28-day intervening interval.

The planned trial duration is 18 months.

Each participant will remain in the trial for 12-13 months, including a screening phase of up to 28 days, intervention phase of 1 day and follow-up phase of 12 months.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 18 years inclusive at time of enrollment and older;
2. Capable to and does provide written informed consent;
3. Able to understand and agrees to comply with planned study procedures and be available for all study visits;
4. Body Mass Index 18-32 kg/square meter, inclusive, at screening;
5. Male or non-pregnant, non-breastfeeding females who agree to comply with applicable contraceptive requirements of the protocol (see Table 1: Acceptable Contraceptive Methods.) Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to initiation of vaccination;
6. Pulse no greater than 100 beats per minute;
7. Systolic blood pressure (BP) is 85 to 150 mmHg, inclusive;
8. Clinical screening laboratory evaluations:

   * Absolute neutrophil count (ANC) ≥1500 cells/mm3
   * Hemoglobin ≥12.0 g/dL for men and ≥11.0 g/dL for women
   * Platelet count ≥120,000/mm3
   * Creatinine clearance (CrCl) >80 mL/min ); Refer to the calculator located on the Frontier Science and Technology Research Foundation (FSTRF) website (at https://www.frontierscience.org/): Calculated Creatinine Clearance - Cockcroft-Gault Equation (Adult).
   * Aspartate aminotransferase (AST) <1.25 x upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) <1.25 x ULN
   * Alkaline phosphatase <2.0 x ULN
   * Total bilirubin <1.1 x ULN
   * Lipase <1.1 x ULN
   * Prothrombin time (PT) <1.1 x ULN
   * Partial thromboplastin time (PTT) <1.1 x ULN
   * CRP < 2.0 x ULN
9. Agree to have samples stored for secondary research related to coronaviruses.

EXCLUSION CRITERIA

1. Positive pregnancy test either at screening or just prior to vaccine administration.
2. Female participant who is breastfeeding or plans to breastfeed from the time of the study vaccination through 3 months after the study vaccination.
3. Has acute or chronic inflammatory condition of the gastrointestinal tract including, but not limited to, Crohn's disease, ulcerative colitis, gastritis, proctitis, or any other inflammatory bowel disorder.
4. Has any medical disease, history, or behavior that may predispose to more severe COVID-19 infection, including hypertension, diabetes, current vaping and/or smoking, history of chronic smoking within the prior year (average of at least one cigarette per day or more), or body mass index of greater than 32; stable hypertension controlled with a stable dose of medication is permitted.
5. Has any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation (including but not limited to acute, subacute, intermittent or chronic medical disease or condition that would place the participant at an unacceptable risk of injury, render the participant unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the participant's successful completion of this trial.)
6. Presence of self-reported or medically documented significant medical or psychiatric condition(s).

   Significant medical or psychiatric conditions include but are not limited to:
   * Respiratory disease (e.g., chronic obstructive pulmonary disease, asthma) requiring daily medications currently or any treatment of respiratory disease exacerbations (e.g., asthma exacerbation) in the last 5 years.
   * Excluded asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics.
   * Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   * Neurological or neurodevelopmental conditions (e.g., migraines, epilepsy, stroke, seizures in the last 3 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis or transverse myelitis).Ongoing malignancy or recent diagnosis of malignancy in the last five years excluding basal cell and squamous cell carcinoma of the skin, which are allowed.
   * An autoimmune disease, including hypothyroidism without a defined non-autoimmune cause, localized or history of psoriasis.
   * An immunodeficiency of any cause or are immune-suppressed.
7. Has an acute illness, as determined by the site PI or appropriate sub-investigator, with or without fever (oral temperature >38.0 degrees Celsius [100.4 degrees Fahrenheit]) within 72 hours prior to study vaccination administration.
8. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
9. Has participated in another investigational study involving any investigational product (study drug, biologic or device) within 60 days, or 5 half-lives, whichever is longer, before study vaccine administration.
10. Currently enrolled in or plans to participate in another clinical trial with an investigational agent (including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) that will be received during the trial period.
11. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
12. Chronic use (more than 14 continuous days) or anticipated use within the next 6 months of any medications that may be associated with impaired immune responsiveness. Including, but not limited to the following excluded drugs: systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1). The use of low dose topical, ophthalmic, inhaled and intranasal steroid preparations will be permitted.
13. Received immunoglobulins and/or any blood or blood products within the 4 months before study vaccine administration or at any time during the study.
14. Has any blood dyscrasias or significant disorder of coagulation.
15. Has any chronic liver disease, including fatty liver.
16. Has a history of alcohol or drug abuse or tests positive for drugs of abuse at screening.
17. Received or plans to receive a licensed, live vaccine within 4 weeks before or after each vaccination.
18. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after each vaccination.
19. Receipt of any other SARS-CoV-2/COVID-19, or other experimental coronavirus vaccine at any time prior to or during the study.
20. Known current or previous laboratory-confirmed SARS CoV-1 OR SARS-CoV-2/COVID-19 infection as documented by a positive PCR test from a nasal swab.
21. Known close contact of anyone with laboratory-confirmed SARS-CoV-2/COVID-19 infection within 2 weeks prior to vaccine administration.
22. Has traveled outside Australia for any duration within 30 days before study vaccination.
23. Currently working in occupation with high risk of exposure to SARS-CoV-2 (e.g., health care worker, emergency response personnel).
24. Allergy to BOTH amoxicillin (or any penicillin derivative) AND erythromycin
25. Household contact, including neonates up to the age of 28 days, with any medical condition or taking medications that may result in immunosuppression.
26. The participant must agree to refrain from donating blood or plasma during the study.
27. Excluded medications (summarized): Excluded asthma medications: inhaled, oral, or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics; Excluded immunosuppressive drugs: systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other similar or toxic drugs during the preceding 6-month period prior to vaccine administration (Day 1); Excluded other medications - current use of any antibiotics, probiotic supplements, H2 blockers or proton pump inhibitors within 7 days prior to vaccination and any anticipated use for 7 days post vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events | Up to12 months post-vaccination
  Adverse events (specifically including incidence of gastrointestinal-associated events) following administration of oral bacTRL-Spike

SECONDARY OUTCOMES:
Immune response against SARS-CoV-2 Spike protein | Baseline (pre-vaccination), and 1, 3 and 12 months post-vaccination
  Antibody against SARS-CoV-2 Spike protein
Incidence of COVID-19 infection | Up to 12 months post-vaccination
  Incidence and clinical phenotype of confirmed and probable COVID-19 infection among vaccinated participants, based on current public health definitions
bacTRL-Spike in stool post-vaccination | Days 8, 15, 22, and 1 and 3 months post-vaccination
  Isolation of viable bacTRL-Spike from stool post-vaccination
Immunity against SARS-CoV-2 | Up to 12 months post-vaccination
  Collection of biological samples for future studies to understand immunity against SARS-CoV-2.

CONTACTS AND LOCATIONS:
Overall Officials: Eric L Sievers, MD, Study Director — Chief Medical Officer; Paul Griffin, FRACP FRCPA FACTM FIML AFACHSM, Principal Investigator — Principal Investigator
Locations (1):
- Nucleus Network Pty Ltd Brisbane (QPharm), Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Undecided